CLINICAL TRIAL: NCT02082795
Title: Investigating Women's Views on the Management of a Breech Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: breechqualyv1
Record Dates: First submitted 2014-03-05; First posted 2014-03-10 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Presentation; Breech, Complicating Pregnancy
Keywords: Breech presentation; External cephalic version; Anaesthesia; Qualitative; Pregnancy
MeSH Terms: conditions — Pregnancy Complications; Breech Presentation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators aim to perform a qualitative study to explore the views of women with a breech presentation on their management in general, and the use of anaesthesia or analgesia for ECV in particular.

DETAILED DESCRIPTION:
Background

Women undergo external cephalic version (ECV) in order to turn a baby in a breech (bottom, or feet down) presentation to a head down position. The procedure traditionally has about a 40% success rate and may be painful, issues that recent literature suggests puts some women off.

Pain relief using a short acting morphine-like painkiller, called remifentanil, can significantly reduce the pain experienced but does not seem to improve ECV success rates. Alternatively, a spinal anaesthetic (similar to that used for a caesarean section) can be used. This increases success rates to around 60% and very effectively reduces pain; however, it is an invasive procedure with potential complications and requires a hospital stay of at least half a day.

Aims and objectives

The investigators aim to perform a qualitative study to explore the views of women with a breech presentation on their management in general, and the use of anaesthesia or analgesia for ECV in particular.

Methods

The investigators will use a semi-structured interview to explore the views of 10-15 expectant mothers recruited from the Breech Clinic at Chelsea and Westminster Hospital. Interviews will be recorded and then transcribed for thematic analysis by two researchers.

Dissemination of output

To our knowledge, this will be the first report on how women view the use of regional anaesthesia and remifentanil analgesia for ECV. In addition, we will add the views of our patient population to the existing literature concerning the management of ECV in general. The investigators anticipate that this information will be used to plan services and to guide future research.

ELIGIBILITY:
Inclusion Criteria:

* Breech presentation
* eligible for an external cephalic version attempt

Exclusion Criteria:

* Multiple pregnancy
* Previous caesarean section
* English not sufficient to carry out the interview

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women found to have a fetus in a breech presentation at >34 weeks gestation following a presentation scan in Chelsea and Westminster Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Mothers' opinions on anaesthesia for external cephalic version | Immediate
  This is a qualitative study using information gathered during a semi-structured interview. All information will be gathered at the time of the interview. There will be no other followup.

SECONDARY OUTCOMES:
Mothers' opinions on management of breech presentation | Immediate
  This is a qualitative study using information gathered during a semi-structured interview. All information will be gathered at the time of the interview. There will be no other followup.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Yentis, BSc MBBS MD MA, Principal Investigator — Chelsea and Westminster Hospital
Locations (1):
- Chelsea and Westminster Hospital, London, United Kingdom